CLINICAL TRIAL: NCT00839644
Title: Airway Secretion Clearance in Cystic Fibrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High dropout, problems recruiting, and smaller than expected decline in FEV1.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cystic Fibrosis Foundation (Other); American Biosystems (currently Hill-Rom) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0609; ACCURS98A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; Chest Wall Oscillation; drainage, postural; Medication Adherence; patient dropouts
MeSH Terms: conditions — Cystic Fibrosis; Medication Adherence; Patient Dropouts | interventions — Chest Wall Oscillation; 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Active Comparator)
  Interventions: Device: Oscillatory Positive Expiratory Pressure
- 3 (Active Comparator)
  Interventions: Other: PD&P: Postural drainage and percussion
- 1 (Active Comparator)
  Interventions: Device: High frequency chest wall oscillation

INTERVENTIONS:
Device: High frequency chest wall oscillation — Therapy prescribed twce daily for twenty minute sessions. High frequency chest wall oscillation (HFCWO) applies sharp compression pulses via an air-pulse generator and inflatable vest. HFCWO generates transient increases in airflow at low lung volumes, cough-like shear forces, and alterations in the consistency of secretions.
  Other Names: Vest
  Arms: 1
Device: Oscillatory Positive Expiratory Pressure — Therapy was prescribed twice daily for 20 minute sessions and included airway vibration, oscillating PEP, and forced expiratory technique (FET) with coughing.
  Other Names: Flutter Device (Scandipharm, Birmingham, AL)
  Arms: 2
Other: PD&P: Postural drainage and percussion — Each of the six positions are to be clapped or vibrated for 4 minutes. After each position the patient is to do three forced expiratory techniques (FET) and cough, continue with FET and coughing until all mobilized mucus has been cleared.
  Other Names: CPT
  Arms: 3

SUMMARY:
The purpose of this study is to compare the effect of three airway secretion clearance techniques (chest physical therapy, flutter device and high frequency chest wall oscillation) on decline in pulmonary function over a three year period in patients with cystic fibrosis.

DETAILED DESCRIPTION:
Study Design: Randomized clinical trial with pulmonary function testing obtained every three months in each of the three treatment groups. Change in slope of FEV1 will be compared. Days of hospitalization and use of oral or IV antibiotics for respiratory tract infection, quality of life, subject satisfaction, and compliance will also be compared.

Sample Size: Enrollment will be completed after 180 subjects have been recruited. Fifteen CF centers will participate.

Subject Selection: Subjects must have the diagnosis of CF, be > 7 years of age and have an FEV1 > 45% of predicted.

Prescribed Therapy: Each subject will receive airway secretion clearance twice a day.

Outcomes: Change in slope of FEV1; days of hospitalization and use of oral or IV antibiotics for respiratory tract infection; quality of life; subject satisfaction; compliance.

ELIGIBILITY:
Inclusion Criteria:

* A proven diagnosis of CF as evidenced by a positive sweat test (as documented by a sweat chloride >60 mEq/L by quantitative pilocarpine iontophoresis), or by the presence of two known CF mutations.
* Aged 7 or older.
* FEV1 >45% (Knudson).
* Able to perform reproducible maneuvers for spirometry at screening as defined by the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines.
* Willing to participate in and comply with the study procedures, and willingness of a parent or legally authorized representative to provide written informed consent.

Exclusion Criteria:

* Hospitalization for complications of CF, or a respiratory exacerbation resulting in - treatment with IV antibiotics within 60 days prior to screening.
* Use of any investigational drug or device within 60 days prior to screening.
* An episode of gross hemoptysis (>249 ml) within 60 days prior to screening, or during the course of the study.
* A pneumothorax in the six months preceding the study or during the course of the study.
* Patients who are pregnant or become pregnant.
* Patients colonized with Burkholderia cepacia.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 1999-12; Primary Completion 2002-12 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
rate of forced expiratory volume in 1 second (FEV1) decline | 3 years

SECONDARY OUTCOMES:
time to need for intravenous (IV) antibiotics to treat pulmonary exacerbations | 3 years
use of other pulmonary therapies | 3 years
adherence to therapy | 3 years
patient satisfaction | 3 years
health-related quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Accurso, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver and The Children's Hospital, Denver, Colorado, United States